CLINICAL TRIAL: NCT02574065
Title: Effects on Crying Time in Colicky Infants With the Supplementation of Lactobacillus Reuteri DSM 17938: A Randomized, Double Blind, Placebo-controlled Study
Brief Title: Effects on Crying Time in Colicky Infants With the Supplementation of Lactobacillus Reuteri DSM 17938
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Children's Hospital (Other)
Collaborators: BioGaia AB (Industry); Suzhou University Affiliated Children's Hospital (Other); Shanghai Children's Medical Center (Other)
Responsible Party: Principal Investigator, Zhang Ting, MD, Shanghai Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSUB0090
Record Dates: First submitted 2015-08-20; First posted 2015-10-12 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Crying Time in Colicky Infants
Keywords: crying; colicky; infants; Lactobacillus reuteri DSM 17938
MeSH Terms: conditions — Crying

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- L. reuteri DSM 17938 group (Experimental): L. reuteri DSM 17938 will be given at a dose of 100000000 colony forming units (CFU) per day in an oil formulation delivered from a drop bottle. In the active study product, freeze-dried L. reuteri is suspended in a mixture of pharmaceutical grade medium chain triglycerides and sunflower oil together with pharmaceutical grade silicon dioxide to give the product the correct rheological properties.
  Each day, at about the same time, the infants will be given 5 drops (1x100000000 CFU) of the study product in connection with feeding.
  Interventions: Drug: L. reuteri DSM 17938
- Placebo group (Placebo Comparator): The placebo consists of an identical formulation without L. reuteri. Each day, at about the same time, the infants will be given 5 drops placebo in connection with feeding.
  Interventions: Other: The placebo consists of an identical formulation without L. reuteri DSM 17938

INTERVENTIONS:
Drug: L. reuteri DSM 17938 — Effects on crying time in colicky infants with the supplementation of Lactobacillus reuteri DSM 17938
  Arms: L. reuteri DSM 17938 group
Other: The placebo consists of an identical formulation without L. reuteri DSM 17938
  Arms: Placebo group

SUMMARY:
Infant colic is a common condition characterized by excessive crying. The otherwise healthy infant aged less than 3 months is difficult to console during the periods with crying. The condition is defined by modified Wessel's criteria i.e. crying for more than 3 hours of the day, for more than 3 days of the week for at least 1 week.

The description of infant colic hasalso been defined by Rome III diagnostic criteria andincludes infants from birth to 4 months of age,without failure to thrive, that are showing paroxysms of irritability, fussing or crying that starts and stops without obvious cause. The episodes last 3 or more hours/day and occur at least 3days/week for at least one week. The infant has no signs of central nervous system or intrinsic developmental difficulties, is normal on physical examination, and has normal growth patterns.

Although infant colic is considered to be self limiting it is a distressing problem for families. It is in fact one of the most common reasons why parents seek the advice of a paediatrician or family practitioner during their child's first 3 months of life Up to 20% of infants under three months are affected by infant colic.

Infant colic could have significant adverse effects on family quality of life and could even be a trigger for shaken baby syndrome. Parental perception associated with colicky complaints is therefor strongly recommended to be an outcome measure in trials of infantile colic.

Measurement of parental/family quality of life and parental perception of colic severity with the help of a Visual Analogue Scale (VAS) in a Polish study showed that the use of a probiotic, Lactobacillus reuteri DSM 17938, could improve the perceived problems.

The relationship between infant colic and gastroenterological, allergical and psychological disorders later in childhood was studied in a prospective study on 96 infants divided into two groups, colicky and non-colicky. The children diagnosed with infant colic, showed an increased susceptibility to recurrent abdominal pain, allergic and psychological disorders in childhood when they were 10 years old.

The aetiology of infantile colic seems to be multifactorialbut is,despite many years of research, still unknown. The intestinal microbiota differs between infants with and without colic and has therefore been suggested to have a potential role. Other possible explanations are for example gut motility disturbances, low-grade mucosal inflammation and visceral hypersensitivity.

Evidence suggests thatadministration of the probioticL. reuteri DSM 17938 might offer some benefit.L. reuteri DSM 17938 has been tested for its effect on crying in colicky infants and has been demonstrated to have a significantly favourable effect on crying time in fivetrials. One is a randomized trial that compared the probioticto Simethicone; three areplacebo controlled randomized double blind trials and yet another is a placebo controlled randomized, single blind, observational study. A fifth studydid not find any effect.

Combining the results in a meta-analysis from three double blind, placebo controlled randomized trials (published at the time of the analysis, including the neutral one) found that, compared with placebo, L. reuteri administration reduced crying time at day 21 with about 40 min.

Recently it has been documented in a clinical trial that prophylactic use of L. reuteriDSM 17938during the first three months of lifereduced the onset offunctional gastrointestinal disorders, particularly functional constipation, regurgitation and infantile colic.

In conclusion, the administration L. reuteri DSM 17938 may reduce the crying time in children with infantile colic, especially those fed predominantly or exclusively with breast milk. However, further randomized controlled studies, are required to be able develop recommendations in the management of infant colic.

The present trial is undertaken to further document the effect of L. reuteri DSM 17938 on crying in colicky infants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis according to modified Wessel's definition of infant colic i.e. crying for more than 3 hours of the day, for more than3 days of the week
* Full term infant, i.e. gestational age between 37 and 42 weeks
* Breast fed, either exclusively or predominantly, i.e. to more than 50%
* Birth weight 2500 - 4000g.
* Apgar score ≥7 at 5 minutes at birth
* Age from birth to 4 months of age
* Parent(s) willingness to postpone major changes in the infant feeding mode
* Parent(s) willingness and ability to fill in diary and questionnaires
* Written informed consent from parents
* Stated availability throughout the study period

Exclusion Criteria:

* Chronic illness or major medical problem
* Gastrointestinal disease
* Failure to thrive
* Use of antibiotics two weeks before randomisation and throughout the intervention period, both infant and mother
* Use of probiotics two weeks before randomisation and throughout the intervention period, both infant (infant formula and/or supplementation)and mother
* Use of proton pump inhibitors two weeks before randomisation and throughout the intervention period.
* Infant receiving solid foods, such as cereals, mashed fruits or vegetable puree
* Participation in other clinical trials

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Daily crying time will be measured at Day 7 through questionnaire finished by parents. | Day 7
  50 evaluable infants in each group will be needed to detect (i.e. get a two-sided p-value less than 5%) a 50 minutes difference in crying time between L. reuteri DSM 17938 and placebo group and with a 90 minutes standard deviation, and a power of 80%, two-sided hypothesis.
Daily crying time will be measured at Day 14 through questionnaire finished by parents. | Day 14
  50 evaluable infants in each group will be needed to detect (i.e. get a two-sided p-value less than 5%) a 50 minutes difference in crying time between L. reuteri DSM 17938 and placebo group and with a 90 minutes standard deviation, and a power of 80%, two-sided hypothesis.
Daily crying time will be measured at Day 21 through questionnaire finished by parents. | Day 21
  50 evaluable infants in each group will be needed to detect (i.e. get a two-sided p-value less than 5%) a 50 minutes difference in crying time between L. reuteri DSM 17938 and placebo group and with a 90 minutes standard deviation, and a power of 80%, two-sided hypothesis.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Zhang, MD, Principal Investigator — Shanghai Children's Hospital
Locations (1):
- Children's Hospital of Shanghai, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Abrahamsson TR, Jakobsson T, Bottcher MF, Fredrikson M, Jenmalm MC, Bjorksten B, Oldaeus G. Probiotics in prevention of IgE-associated eczema: a double-blind, randomized, placebo-controlled trial. J Allergy Clin Immunol. 2007 May;119(5):1174-80. doi: 10.1016/j.jaci.2007.01.007. Epub 2007 Mar 8. PMID 17349686
- [Background] Barr RG, Kramer MS, Boisjoly C, McVey-White L, Pless IB. Parental diary of infant cry and fuss behaviour. Arch Dis Child. 1988 Apr;63(4):380-7. doi: 10.1136/adc.63.4.380. PMID 3365007
- [Background] Chau K, Lau E, Greenberg S, Jacobson S, Yazdani-Brojeni P, Verma N, Koren G. Probiotics for infantile colic: a randomized, double-blind, placebo-controlled trial investigating Lactobacillus reuteri DSM 17938. J Pediatr. 2015 Jan;166(1):74-8. doi: 10.1016/j.jpeds.2014.09.020. Epub 2014 Oct 23. PMID 25444531
- [Background] Hyman PE, Milla PJ, Benninga MA, Davidson GP, Fleisher DF, Taminiau J. Childhood functional gastrointestinal disorders: neonate/toddler. Gastroenterology. 2006 Apr;130(5):1519-26. doi: 10.1053/j.gastro.2005.11.065. PMID 16678565
- [Background] Indrio F, Riezzo G, Raimondi F, Bisceglia M, Cavallo L, Francavilla R. The effects of probiotics on feeding tolerance, bowel habits, and gastrointestinal motility in preterm newborns. J Pediatr. 2008 Jun;152(6):801-6. doi: 10.1016/j.jpeds.2007.11.005. Epub 2007 Dec 26. PMID 18492520
- [Background] Indrio F, Di Mauro A, Riezzo G. Prophylactic use of a probiotic in the prevention of colic, regurgitation, and functional constipation--reply. JAMA Pediatr. 2014 Aug;168(8):778. doi: 10.1001/jamapediatrics.2014.368. No abstract available. PMID 25090301
- [Background] Lucassen PL, Assendelft WJ, van Eijk JT, Gubbels JW, Douwes AC, van Geldrop WJ. Systematic review of the occurrence of infantile colic in the community. Arch Dis Child. 2001 May;84(5):398-403. doi: 10.1136/adc.84.5.398. PMID 11316682
- [Background] Savino F, Cresi F, Pautasso S, Palumeri E, Tullio V, Roana J, Silvestro L, Oggero R. Intestinal microflora in breastfed colicky and non-colicky infants. Acta Paediatr. 2004 Jun;93(6):825-9. PMID 15244234
- [Background] Savino F, Bailo E, Oggero R, Tullio V, Roana J, Carlone N, Cuffini AM, Silvestro L. Bacterial counts of intestinal Lactobacillus species in infants with colic. Pediatr Allergy Immunol. 2005 Feb;16(1):72-5. doi: 10.1111/j.1399-3038.2005.00207.x. PMID 15693915
- [Background] Savino F, Pelle E, Palumeri E, Oggero R, Miniero R. Lactobacillus reuteri (American Type Culture Collection Strain 55730) versus simethicone in the treatment of infantile colic: a prospective randomized study. Pediatrics. 2007 Jan;119(1):e124-30. doi: 10.1542/peds.2006-1222. PMID 17200238
- [Background] Steutel NF, Benninga MA, Langendam MW, de Kruijff I, Tabbers MM. Reporting outcome measures in trials of infant colic. J Pediatr Gastroenterol Nutr. 2014 Sep;59(3):341-6. doi: 10.1097/MPG.0000000000000412. PMID 24796800
- [Background] Sung V, Hiscock H, Tang ML, Mensah FK, Nation ML, Satzke C, Heine RG, Stock A, Barr RG, Wake M. Treating infant colic with the probiotic Lactobacillus reuteri: double blind, placebo controlled randomised trial. BMJ. 2014 Apr 1;348:g2107. doi: 10.1136/bmj.g2107. PMID 24690625
- [Background] Szajewska H, Gyrczuk E, Horvath A. Lactobacillus reuteri DSM 17938 for the management of infantile colic in breastfed infants: a randomized, double-blind, placebo-controlled trial. J Pediatr. 2013 Feb;162(2):257-62. doi: 10.1016/j.jpeds.2012.08.004. Epub 2012 Sep 14. PMID 22981952
- [Background] de Weerth C, Fuentes S, Puylaert P, de Vos WM. Intestinal microbiota of infants with colic: development and specific signatures. Pediatrics. 2013 Feb;131(2):e550-8. doi: 10.1542/peds.2012-1449. Epub 2013 Jan 14. PMID 23319531
- [Background] WESSEL MA, COBB JC, JACKSON EB, HARRIS GS Jr, DETWILER AC. Paroxysmal fussing in infancy, sometimes called colic. Pediatrics. 1954 Nov;14(5):421-35. No abstract available. PMID 13214956